CLINICAL TRIAL: NCT04295538
Title: A Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Assess the Safety and Efficacy of Elezanumab in Acute Traumatic Cervical Spinal Cord Injury
Brief Title: Safety And Efficacy Study Of Intravenous (IV) Administration Of Elezanumab To Assess Change In Upper Extremity Motor Score (UEMS) In Adult Participants With Acute Traumatic Cervical Spinal Cord Injury (SCI)
Acronym: ELASCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-077; 2019-003752-36 (EudraCT Number)
Expanded Access: NCT04278235 (Available)
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Spinal Cord Injury (SCI); Cervical Spinal Cord Injury; Cervical SCI; Elezanumab; ABT-555; Upper Extremity Motor Score (UEMS); Acute Traumatic Cervical Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — elezanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo for elezanumab
  Interventions: Drug: Placebo
- Elezanumab (Experimental): Participants will receive elezanumab dose A
  Interventions: Drug: Elezanumab

INTERVENTIONS:
Drug: Elezanumab — Solution for infusion; Intravenous (IV)
  Other Names: ABT-555
  Arms: Elezanumab
Drug: Placebo — Solution for infusion; Intravenous (IV)
  Arms: Placebo

SUMMARY:
Acute Spinal Cord Injury (SCI) is a rare injury that leads to permanent neuromotor impairment and sudden disability. Approximately 25,000 people experience cervical SCI in the United States, Europe, and Japan every year. The purpose of this study is to see if elezanumab is safe and assess change in Upper Extremity Motor Score (UEMS) in participants with acute traumatic cervical SCI.

Elezanumab is an investigational drug being developed for the treatment of SCI. Elezanumab is a monoclonal antibody, that binds to an inhibitor of neuronal regeneration and neutralizes the inhibitor, thus potentially promoting neuroregeneration. This study is "double-blinded", which means that neither trial participants nor the study doctors will know who will be given which study drug. Study doctors put the participants in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to placebo. Participants 18-75 years of age with a SCI will be enrolled. Approximately 54 participants will be enrolled in the study in approximately 49 sites worldwide.

Participants will receive intravenous (IV) doses of elezanumab or placebo within 24 hours of injury and every 4 weeks thereafter through Week 48 for a total of 13 doses.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic cervical spinal cord injury (SCI), neurological level of injury of C4, C5, C6, or C7 with no damage to cord in thoracic (T2 and beyond) and lumbar regions that, in the investigator's opinion, would significantly limit recovery.
* Maximum screening UEMS of 32.
* American Spinal Injury Association Impairment Scale (AIS) grade A or B at Screening.
* Able to initiate study drug administration within 24 hours of injury.
* Participants with comorbid conditions that, in the investigator's opinion, are clinically stable and not expected to meaningfully progress in the following 12 months, may be considered eligible to participate.

Exclusion Criteria:

* Evidence of complete spinal cord transection.
* Significant concomitant head injury with a clinically significant abnormality on a head computed tomography (CT).
* One or more upper extremity muscle groups untestable (e.g., immobilized or restricted by a cast) during the screening International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) examination.
* Known receipt of any other investigational product within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
* Female who is pregnant, breastfeeding, or considering becoming pregnant during the study or for within 39 weeks (5 half-lives) after the last dose of study drug.
* The cause of the acute SCI is one of the following: from gunshot or penetrating/stab wound; non-traumatic SCI, results of seizure, or known attempted suicide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-06 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Motor Score (UEMS) | 52 Weeks
  The UEMS is a subscore of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) that grades function of 5 key muscles in the upper limbs on a scale of 0 to 5 on each side from total paralysis to active full range of movement, respectively.
Number of Participants Experiencing Adverse Events | Up to approximately 91 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in Spinal Cord Independence Measures (SCIM III) Self-Care Score | Week 0 through Week 52
  The SCIM III self-care score addresses four areas of self-care management: feeding, grooming, bathing, and dressing. It has a total of 4 questions. Scores range from 0-20 where a score of 0 defines total dependence and 20 is indicative of complete independence.
Change in Upper Extremity Motor Score (UEMS) From Baseline | Week 0 through Week 52
  The UEMS is a subscore of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) that grades function of 5 key muscles in the upper limbs on a scale of 0 to 5 on each side from total paralysis to active full range of movement, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (22):
  - University of California Davis Health /ID# 224892, Sacramento, California
  - Shepherd Center, Inc /ID# 230370, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 218009, Chicago, Illinois
  - University of Louisville Hospital /ID# 215948, Louisville, Kentucky
  - Duplicate_Tufts Medical Center /ID# 225410, Boston, Massachusetts
  - Brigham & Women's Hospital /ID# 216342, Boston, Massachusetts
  - Duplicate_Boston University School of Medicine /ID# 218371, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 218149, Boston, Massachusetts
  - Regents of the University of Michigan /ID# 215890, Ann Arbor, Michigan
  - Washington University-School of Medicine /ID# 215325, St Louis, Missouri
  - Hackensack Univ Med Ctr /ID# 215754, Hackensack, New Jersey
  - Jersey Shore University Medical Center /ID# 218162, Neptune City, New Jersey
  - Rutgers New Jersey School of Medicine /ID# 216212, Newark, New Jersey
  - Duplicate_Duke Cancer Center /ID# 216888, Durham, North Carolina
  - Oregon Medical Research Center /ID# 227371, Portland, Oregon
  - University of Pennsylvania /ID# 218662, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 215460, Philadelphia, Pennsylvania
  - University of Virginia Health /ID# 218117, Charlottesville, Virginia
  - Sentara Norfolk General Hospital /ID# 218302, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 217481, Richmond, Virginia
  - West Virginia University Hospitals /ID# 217344, Morgantown, West Virginia
  - Wisconsin Medical Center /ID# 215610, Milwaukee, Wisconsin
- Royal Adelaide Hospital /ID# 216953, Adelaide, South Australia, Australia
- Canada (5):
  - Foothills Medical Centre /ID# 214790, Calgary, Alberta
  - QEII - Health Sciences Centre /ID# 215249, Halifax, Nova Scotia
  - The Ottawa Hospital Civic Campus /ID# 215270, Ottawa, Ontario
  - Toronto Western Hospital /ID# 215214, Toronto, Ontario
  - CIUSSS du Nord-de-l'ile-de-Montréal_Hopital du Sacré-Coeur de Montréal /ID# 215210, Montreal, Quebec
- The Chaim Sheba Medical Center /ID# 240917, Ramat Gan, Tel Aviv, Israel
- Japan (4):
  - NHO Nagoya Medical Center /ID# 239617, Nagoya, Aichi-ken
  - Funabashi Municipal Medical Center /ID# 225599, Funabashi-shi, Chiba
  - Japan Organization of Occupational Health and Safety Spinal Injuries Centre /ID# 224141, Iizuka-shi, Fukuoka
  - National Hospital Organization Murayama Medical Center /ID# 223492, Musashimurayama-shi, Tokyo
- South Korea (2):
  - Ajou University Hospital /ID# 241119, Suwon, Gyeonggido
  - Duplicate_Inha University Hospital /ID# 238890, Junggu, Incheon Gwang Yeogsi
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña /ID# 216384, A Coruña, A Coruna
  - Hospital Universitario Vall de Hebron /ID# 217794, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 225354, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 225692, Seville
  - Hospital Nacional de Paraplejicos /ID# 225508, Toledo
  - Hospital Universitario y Politecnico La Fe /ID# 217797, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/